CLINICAL TRIAL: NCT04999176
Title: A Multicenter, Open-label, Prospective, Randomized, Active-controlled Study on the Efficacy and Safety of Oral Rivaroxaban Versus Enoxaparin for Venous Thromboembolism Prophylaxis After Major Gynecological Cancer Surgery.
Brief Title: Venous Thromboembolism Prophylaxis After Gynecological Pelvic Cancer Surgery With Rivaroxaban vs Enoxaparin
Acronym: VALERIA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: André Luiz Malavasi Longo de Oliveira (Other)
Collaborators: Science Valley Research Institute (Other)
Responsible Party: Sponsor-Investigator, André Luiz Malavasi Longo de Oliveira, Clinical Director - São Paulo State Public Women's Health Reference Center, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VALERIA TRIAL
Record Dates: First submitted 2021-08-03; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Cancer; Rivaroxaban; Venous Thromboembolism; Thromboprophylaxis
Keywords: Direct oral anticoagulants; Gynecologic cancer; Low-molecular weight heparin
MeSH Terms: conditions — Neoplasms; Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Intervention Model Description: This study aims to evaluate the efficacy and safety of oral rivaroxaban 10 mg for 30 days in thromboprophylaxis after gynecological pelvic cancer surgery compared to subcutaneous enoxaparin 40 mg. The primary efficacy outcome is a combination of symptomatic VTE and VTE-related death or VTE detected by mandatory Doppler ultrasound on day 30±4 post-operative. The primary safety outcome is the incidence of major and clinically relevant non-major bleeding according to ISTH criteria.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban (Experimental): Oral Rivaroxaban (10 mg once daily) for 30 days post-operative
  Interventions: Drug: Rivaroxaban
- Enoxaparin (Active Comparator): Subcutaneous Enoxaparin (40 mg once daily) for 30 days post-operative
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban — Patients will be submitted to an initial screening evaluation during hospitalization. At discharge, they will be randomized and enrolled to be treated with oral rivaroxaban (10 mg once daily, for 30 days), once randomized to this group. A mandatory lower limb Doppler ultrasound will be carried out on day 30±4 as part of the primary efficacy endpoint. A final follow-up phone call visit will be performed on day 60 postoperative.
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Enoxaparin — Patients will be submitted to an initial screening evaluation during hospitalization. At discharge, they will be randomized and enrolled to be treated with subcutaneous enoxaparin (40 mg once daily, for 30 days), once randomized to this group. A mandatory lower limb Doppler ultrasound will be carried out on day 30±4 as part of the primary efficacy endpoint. A final follow-up phone call visit will be performed on day 60 postoperative.
  Other Names: Clexane
  Arms: Enoxaparin

SUMMARY:
The Valeria trial will provide high-quality evidence regarding the efficacy and safety of oral rivaroxaban in thromboprophylaxis after gynecological pelvic cancer surgery in comparison with standard parenteral enoxaparin.

DETAILED DESCRIPTION:
Cancer-associated thrombosis is the second leading cause of mortality in cancer patients, mainly due to the most common complication, venous thromboembolism (VTE). New oral antithrombotic strategies for VTE prevention after gynecological cancer surgery might be non-inferior to parenteral low-molecular-weight heparin (LMWH) in efficacy and safety with increased adherence, comfort, and reduced costs.

This is a multicenter, open-label, prospective, randomized, active-controlled study, and non-inferiority trial. Four hundred and forty patients submitted to major gynecological cancer surgery will be randomized in a 1:1 ratio to receive either oral rivaroxaban 10 mg once daily or subcutaneous enoxaparin 40mg once daily for 30 days post-operative. The primary efficacy outcome is a combination of symptomatic VTE and VTE-related death or VTE detected by mandatory Doppler ultrasound on day 30±4 post-operative. The primary safety outcome is the incidence of major and clinically relevant non-major bleeding according to the International Society on Thrombosis and Hemostasis criteria.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years of age or older
* Have undergone major gynecological cancer surgery (staging surgery, debulking surgery, -
* Total or radical hysterectomy, unilateral or bilateral salpingo-oophorectomy, omentectomy, lymph node removal, open or laparoscopic access)
* Have signed informed consent
* Have received thromboprophylaxis with low-molecular-weight heparin, fondaparinux, or unfractionated heparin during the index hospitalization

Exclusion Criteria:

* Age < 18 years
* Refusal of informed consent
* Physician decision that involvement in the trial was not in the patient's best interest
* Patients with a medical indication for anticoagulation therapy at the time of inclusion (for example, diagnosis of venous thromboembolism, atrial fibrillation, mechanical valve prosthesis)
* Patients with contraindications to anticoagulation (active bleeding, liver failure, blood dyscrasia, or prohibitive hemorrhagic risk in the investigator's assessment)
* Active cancer (excluding non-melanoma skin cancer) defined as cancer not in remission or radiotherapy requiring active chemotherapy or adjunctive therapies such as immunotherapy
* Use of strong inhibitors of cytochrome P450 (CYP) 3A4 and/or glycoprotein P (P-gp) (eg, protease inhibitors, ketoconazole, Itraconazole) and/or use of P-gp and strong inducers of CYP3A4 (how but not limiting rifampicin/rifampicin, rifabutin, rifapentine, phenytoin, phenobarbital, carbamazepine or St. John's wort)
* Creatinine clearance <30 ml / min
* Pregnancy or breastfeeding
* Known HIV infection
* Presence of one of the following uncontrolled or unstable cardiovascular diseases: stroke, ECG confirmed acute ischemia or myocardial infarction, and/or clinically significant dysrhythmia

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2020-10-22 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Venous thromboembolism and VTE related-death | At day 30 +/- post hospital discharge
  A composite of symptomatic objectively confirmed VTE (deep venous thrombosis, pulmonary embolism, and asymptomatic ultrasonography-confirmed, deep venous thrombosis or venous thromboembolism-related death at 30 days post-operative.

SECONDARY OUTCOMES:
Clinically relevant bleeding | At day 30 +/- post hospital discharge
  A combination of major bleeding plus clinically relevant non-major bleeding at 30 days post-operative.

OTHER OUTCOMES:
A composite of myocardial infarction, stroke, arrhythmias, heart failure, venous thromboembolism (VTE), and all-cause death | At day 30 +/- post hospital discharge
  A composite of myocardial infarction, stroke, arrhythmias, heart failure, venous thromboembolism (VTE), and all-cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Ramacciotti, MD, PhD, Study Chair — Science Valley Research Institute
Locations (1):
- Science Valley Research Institute, Santo André, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohashi Y, Ikeda M, Kunitoh H, Sasako M, Okusaka T, Mukai H, Fujiwara K, Nakamura M, Kimura T, Ibusuki K, Sakon M. Venous thromboembolism in patients with cancer: design and rationale of a multicentre, prospective registry (Cancer-VTE Registry). BMJ Open. 2018 May 30;8(5):e018910. doi: 10.1136/bmjopen-2017-018910. PMID 29848769
- [Background] Comerota AJ, Ramacciotti E. A Comprehensive Overview of Direct Oral Anticoagulants for the Management of Venous Thromboembolism. Am J Med Sci. 2016 Jul;352(1):92-106. doi: 10.1016/j.amjms.2016.03.018. Epub 2016 Apr 6. PMID 27432042
- [Background] Guntupalli SR, Brennecke A, Behbakht K, Tayebnejad A, Breed CA, Babayan LM, Cheng G, Ramzan AA, Wheeler LJ, Corr BR, Lefkowits C, Sheeder J, Matsuo K, Flink D. Safety and Efficacy of Apixaban vs Enoxaparin for Preventing Postoperative Venous Thromboembolism in Women Undergoing Surgery for Gynecologic Malignant Neoplasm: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e207410. doi: 10.1001/jamanetworkopen.2020.7410. PMID 32589230
- [Background] Key NS, Khorana AA, Kuderer NM, Bohlke K, Lee AYY, Arcelus JI, Wong SL, Balaban EP, Flowers CR, Francis CW, Gates LE, Kakkar AK, Levine MN, Liebman HA, Tempero MA, Lyman GH, Falanga A. Venous Thromboembolism Prophylaxis and Treatment in Patients With Cancer: ASCO Clinical Practice Guideline Update. J Clin Oncol. 2020 Feb 10;38(5):496-520. doi: 10.1200/JCO.19.01461. Epub 2019 Aug 5. PMID 31381464
- [Background] Chan NC, Weitz JI. Rivaroxaban for prevention and treatment of venous thromboembolism. Future Cardiol. 2019 Mar;15(2):63-77. doi: 10.2217/fca-2018-0076. Epub 2019 Feb 19. PMID 30779598